CLINICAL TRIAL: NCT00249054
Title: Clinical Performance of the ASR and ReCap Resurfacing Implants-7Years Follow-Up.
Brief Title: Prospective Clinical Evaluation of ASR and ReCap Resurfacing Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Arne Borgwardt, Head of Dpt, Frederiksberg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF11279577
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Patients Suitable for THA

ARMS (2):
- ASR hip prosthesis (Active Comparator): DuPuy ASR hip prosthesis
  Interventions: Device: ASR hip prosthesis; Device: ReCap hip prosthesis
- ReCap hip prosthesis (Active Comparator): Biomet ReCap hip prosthesis
  Interventions: Device: ReCap hip prosthesis

INTERVENTIONS:
Device: ASR hip prosthesis — Implantation of resurfacing prosthesis
  Other Names: DuPuy ASR hip prosthesis
  Arms: ASR hip prosthesis
Device: ReCap hip prosthesis — Implantation of resurfacing prosthesis
  Other Names: Biomet ReCap hip prosthesis

SUMMARY:
This evaluation is being conducted to evaluate the performance of the ASR arthroplasty. The performance of the devices will be assessed by:

Clinical parameters: pain, function, satisfaction and complications. Blood samples: Analyse of metal ions, lymphocyte migration, lymphocyte proliferation assay and cytokines.

Biopsies: Metal ions, cytokines and histology. Biomechanics: Strength, gait analysis, range of motion. Scanning: DEXA and MRI

ELIGIBILITY:
Inclusion Criteria:

ASA I-II,DEXA-scanning:

* lower limit for a 55 years old women,
* MRI normal
* vitality in caput
* willing to return for follow-up evaluations.

Exclusion Criteria:

* collum femoris < 2 cm
* large cysts in caput (> 1 cm)
* mismatch between caput and acetabulum
* caput necrosis
* treatment with medicine which affects bone metabolism
* impaired kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-11; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical Performance of the ASR and ReCap Resurfacing Implants-7Years Follow-Up. | 10 year follow up
  follow with intervals of 1 to 3 years for determination of function and prosthesis survival

CONTACTS AND LOCATIONS:
Overall Officials: arne borgwardt, M.D., Study Director — Frederiksberg University Hospital
Locations (1):
- Frederiksberg University Hospital, Frederiksberg, Copenhagen, Denmark